CLINICAL TRIAL: NCT05186376
Title: Accuracy of Maxillary Repositioning With bi or Tripartite Disjonction by Virtual Planning in Orthognathic Surgery Using Patient-specific Titanium Plates : a Case Series
Brief Title: Accuracy of Maxillary Repositioning With bi or Tripartite Disjonction by Virtual Planning in Orthognathic Surgery Using Patient-specific Titanium Plates
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21IUFC02
Record Dates: First submitted 2021-12-27; First posted 2022-01-11 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Occlusal Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: bimaxillair osteotomy with maxillar segmentation — Patients who underwent bimaxillair osteotomy with maxillar segmentation

SUMMARY:
The aim of this study was to assess the accuracy of computer-aided orthognathic surgery and patient specific titanium plates for maxillar osteotomy with bi or tripartite disjonction in 22 patients who underwent bimaxillar osteotomy for occlusal trouble.

ELIGIBILITY:
Inclusion Criteria:

- bimaxillar osteotomy with maxillar segmentation and full imageries .

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 22 patients, who underwent bimaxillar osteotomy with maxillar segmentation, in Nice from September 2017 to July 2021, operated by Charles SAVOLDELLI, using patient-specific implants
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
accuracy of patient-specific surgical guides and plates in maxillary repositioning with bi or tri-partite disjonction | 2 months
  Error (in millimeters) in repositionning the maxilla comaring 3D-plannification skulls and post-operative CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital - IUFC, Nice, France

IPD SHARING:
Plan to Share IPD: No